CLINICAL TRIAL: NCT01608620
Title: The Relation of Total and Individual Fructose-containing Sugars With Incident Cardiometabolic Diseases: A Series of Systematic Reviews and Meta-analyses of Prospective Observational Studies
Brief Title: Meta-analyses of Total and Individual Fructose-containing Sugars and Incident Cardiometabolic Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: Calorie Control Council (Other); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Adjunct Research Fellow, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CCC-Sugars epi 2012
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Overweight; Obesity; Dyslipidemia; Hyperlipidemia; Diabetes; Prediabetes; Dysglycemia; Gout; Hypertension; Metabolic Syndrome; Coronary Heart Disease; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; High fructose corn syrup; Fruit; Isocaloric; Hypercaloric; Cardiometabolic risk factors; Triglycerides; Cholesterol; Glycemic control; Insulin resistance; Body weight; Uric acid; Blood pressure
MeSH Terms: conditions — Overweight; Obesity; Dyslipidemias; Hyperlipidemias; Diabetes Mellitus; Prediabetic State; Gout; Hypertension; Metabolic Syndrome; Coronary Disease; Cardiovascular Diseases; Insulin Resistance; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Since uncontrolled observational studies first linked fructose to the epidemic of obesity almost a decade ago, it has become a focus of intense concern regarding its role in the obesity epidemic and increasing burden of cardiometabolic disease. Despite the uncertainties in the evidence, international health organizations have cautioned against moderate to high intakes fructose-containing sugars, especially those from sugar sweetened beverages (SSBs). To improve the evidence on which nutrition recommendations are based, the investigators propose to study of the role of fructose-containing sugars in the development of overweight/obesity, diabetes, hypertension, gout, and cardiovascular disease, by undertaking a series of systematic syntheses of the available prospective cohort studies. Prospective cohort studies have the advantage of relating "real world" intakes of sugars to clinically meaningful disease endpoints over long durations of follow-up. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing recommendations for the general public, as well as those at risk of diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
Background: Fructose has become a focus of intense concern regarding its links to the obesity epidemic and increasing burden of cardiometabolic disease. There have been dozens of editorials, commentaries, and letters in the scientific literature and numerous pieces in the lay and social media calling for efforts to restrict its intake and even regulate it like tobacco or alcohol. Uncontrolled ecological analyses which have linked increasing fructose intake with increasing obesity, diabetes, and hypertension rates and animal models of fructose induced metabolic syndrome and hypertension, which overfeed fructose at levels of exposure far beyond actual population levels of intake, have been used to underpin this debate. Evidence from well-adjusted prospective cohort studies also suggest a positive association between the consumption of sugar-sweetened beverages and increased energy consumption and weight gain. But not all meta-analyses of the available prospective cohort studies have supported this conclusion for SSBs, and no meta-analyses have investigated the effect of total fructose-containing sugars which also include grain and fruit sources on incident overweight/obesity, diabetes, metabolic syndrome, hypertension, gout, and cardiovascular disease. Despite the limitations in extrapolating from the available observational data and their inconsistency with data from controlled trials in humans (the highest level of evidence used in evidence based medicine) which do not show any adverse metabolic effects under isocaloric feeding conditions, the heart and diabetes associations have taken a risk reduction approach to added fructose-containing sugars, setting highly restrictive upper thresholds for their intake to achieve and maintain healthy body-weights and avoid adverse lipid effects.

Objective: To improve the evidence on which recommendations and public health policy are based, we will conduct a series of systematic reviews and meta-analyses of the role of fructose-containing sugars in the development of cardiometabolic disease in prospective cohort studies. A total of 5 analyses are proposed: (1)overweight/obesity, (2) diabetes/metabolic syndrome, (3) hypertension, (4) gout, and (5) coronary heart disease (CHD).

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Meta-analysis Of Observational Studies in Epidemiology (MOOSE) guidelines.

Data sources. MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms, supplemented by manual, hand searches of bibliographies.

Study selection: We will include prospective cohort studies investigating the relation of fructose-containing (fructose, sucrose, and HFCS) sugars to incident overweight/obesity, diabetes, metabolic syndrome, hypertension, gout, and cardiovascular disease.

Data extraction. Two investigators will independently extract information about study design, sample size, subject characteristics, fructose form, fructose exposure levels, duration/person-years of follow-up, background diet profile, adjustments of models. Risk ratios for clinical outcomes will be extracted or derived from clinical event data across quantiles of exposure. Risk of bias will be assessed using the Cochrane Risk of Bias tool.

Outcomes: Each of the 5 proposed analyses will assess a different cardiometabolic disease outcome: (1) overweight/obesity, (2) diabetes/metabolic syndrome, (3) hypertension, (4) gout, and (5) CHD.

Data synthesis. The natural log-transformed relative risks of clinical outcomes comparing the highest exposure level to the reference group from each cohort will be pooled using the generic inverse variance method with random effects models. Heterogeneity will be assessed by Cochrane's Q and quantified by I2. Sensitivity analyses and a priori subgroup analyses will be undertaken to explore sources of heterogeneity including the effect of underlying disease status, sex, sugar type (fructose, sucrose, HFCS), follow-up (<10-years, >=10-years), level of adjustment of models, and Cochrane risk of bias on the effect of fructose. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses. Meta-regression analyses will assess the significance of subgroups analyses. Dose-response analyses will be undertaken using random-effects generalized least squares trend estimation models (GLST), appropriate for weighted regression of summarized dose-response data with dependent components(i.e. the reference exposure level). If insufficient evidence of a linear relationship is found, then we will do spline curve modeling (the MKSPLINE procedure) to characterize segments of the dose response curve where a linear approximation best describes the data. Publication bias will be assessed by the inspection of funnel plots and using Begg's and Egger's tests.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Preliminary findings: To address the uncertainties in the evidence, we conducted a series of Canadian Institutes of Health Research (CIHR) funded systematic reviews and meta-analyses of controlled feeding trials of the effect of fructose on cardiometabolic risk (ClinicalTrials.gov registration number: NCT01363791). We found that fructose in isocaloric substitution for other sources of carbohydrate (isocaloric trials) does not increase body weight, lipids, blood pressure, uric acid, or insulin and even improves glycemic control. There was, however, a signal for harm under certain conditions. High doses of fructose increased triglycerides in isocaloric trials, and fructose providing excess energy at extreme doses relative to control diets (hypercaloric trials) also increased body weight, triglycerides, and uric acid. The implications of these findings for "real world" dietary advice, however, were complicated by several factors. First, fructose is not commonly consumed in isolation as a sweetener. Sucrose and HFCS are the primary fructose-containing sweeteners in the U.S. diet. Second, the level of fructose exposure in the available trials was well above population levels of intake, exceeding the 95th-percentile for U.S. intake in most of the isocaloric trials and in all of the hypercaloric trials, in which the excess energy brought by fructose was an important source of confounding. Finally, the available trials investigated effects on biomarkers of disease and not clinically meaningful events. The proposed systematic review and meta-analyses of prospective cohort studies will address these limitations directly by investigating the relation of self-reported, "real world" intakes of all fructose-containing sugars (fructose, sucrose, and HFCS) to the development overweight/obesity, diabetes/metabolic syndrome, hypertension, gout, and cardiovascular disease.

Significance: The proposed project will aid in knowledge translation related to the effects of dietary fructose on overweight/obesity, diabetes/metabolic syndrome, hypertension, gout, and cardiovascular disease, strengthening the evidence-base for recommendations and improving health outcomes through informing consumers and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Prospective observational studies
* Assessment of fructose-containing sugar exposure
* Viable clinical outcome data by level of exposure

Exclusion Criteria:

* Ecological, cross-sectional, and retrospective observational studies, clinical trials, and non-human studies
* No assessment of fructose-containing sugar exposure
* No viable clinical outcome data by level of exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Overweight/obesity analysis | up to 1.5-years
  Risk ratios for incident Overweight and obesity by total fructose-containing sugar exposure
Diabetes/metabolic syndrome analysis | Up to 1.5-years
  Risk ratios for incident diabetes and metabolic syndrome by total fructose-containing sugar exposure
Hypertension analsysis | Up to 1.5-years
  Risk ratios for incident hypertension by total fructose-containing sugar exposure
Gout analysis | Up to 1.5-years
  Risk ratios for incident gout by total fructose-containing sugar exposure
Coronary heart disease (CHD) analysis | Up to 1.5-years
  Risk ratios for incident CHD by total fructose-containing sugar exposure

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Study Director — Department of Pathology and Molecular Medicine, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Russell J de Souza, ScD, RD, Study Director — Department of Epidemiology and Biostatistics, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, Carleton AJ, Chatha S, Jiang HY, de Souza RJ, Beyene J, Kendall CW, Jenkins DJ. Heterogeneous effects of fructose on blood lipids in individuals with type 2 diabetes: systematic review and meta-analysis of experimental trials in humans. Diabetes Care. 2009 Oct;32(10):1930-7. doi: 10.2337/dc09-0619. Epub 2009 Jul 10. PMID 19592634
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Chiavaroli L, Wang DD, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Dibuono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Hypertension. 2012 Apr;59(4):787-95. doi: 10.1161/HYPERTENSIONAHA.111.182311. Epub 2012 Feb 13. PMID 22331380
- [Background] Sievenpiper JL, de Souza RJ, Mirrahimi A, Yu ME, Carleton AJ, Beyene J, Chiavaroli L, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. Effect of fructose on body weight in controlled feeding trials: a systematic review and meta-analysis. Ann Intern Med. 2012 Feb 21;156(4):291-304. doi: 10.7326/0003-4819-156-4-201202210-00007. PMID 22351714
- [Background] Wang DD, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. The effects of fructose intake on serum uric acid vary among controlled dietary trials. J Nutr. 2012 May;142(5):916-23. doi: 10.3945/jn.111.151951. Epub 2012 Mar 28. PMID 22457397
- [Background] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Background] Sievenpiper JL, de Souza RJ, Jenkins DJ. Sugar: fruit fructose is still healthy. Nature. 2012 Feb 22;482(7386):470. doi: 10.1038/482470e. No abstract available. PMID 22358823
- [Background] Sievenpiper JL, de Souza RJ, Kendall CW, Jenkins DJ. Is fructose a story of mice but not men? J Am Diet Assoc. 2011 Feb;111(2):219-20; author reply 220-2. doi: 10.1016/j.jada.2010.12.001. No abstract available. PMID 21272692
- [Result] Jayalath VH, Sievenpiper JL, de Souza RJ, Ha V, Mirrahimi A, Santaren ID, Blanco Mejia S, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Total fructose intake and risk of hypertension: a systematic review and meta-analysis of prospective cohorts. J Am Coll Nutr. 2014;33(4):328-39. doi: 10.1080/07315724.2014.916237. Epub 2014 Aug 21. PMID 25144126
- [Derived] Khan TA, Tayyiba M, Agarwal A, Mejia SB, de Souza RJ, Wolever TMS, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Relation of Total Sugars, Sucrose, Fructose, and Added Sugars With the Risk of Cardiovascular Disease: A Systematic Review and Dose-Response Meta-analysis of Prospective Cohort Studies. Mayo Clin Proc. 2019 Dec;94(12):2399-2414. doi: 10.1016/j.mayocp.2019.05.034. PMID 31806098
- [Derived] Tsilas CS, de Souza RJ, Mejia SB, Mirrahimi A, Cozma AI, Jayalath VH, Ha V, Tawfik R, Di Buono M, Jenkins AL, Leiter LA, Wolever TMS, Beyene J, Khan T, Kendall CWC, Jenkins DJA, Sievenpiper JL. Relation of total sugars, fructose and sucrose with incident type 2 diabetes: a systematic review and meta-analysis of prospective cohort studies. CMAJ. 2017 May 23;189(20):E711-E720. doi: 10.1503/cmaj.160706. PMID 28536126
- [Derived] Jamnik J, Rehman S, Blanco Mejia S, de Souza RJ, Khan TA, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ, Sievenpiper JL. Fructose intake and risk of gout and hyperuricemia: a systematic review and meta-analysis of prospective cohort studies. BMJ Open. 2016 Oct 3;6(10):e013191. doi: 10.1136/bmjopen-2016-013191. PMID 27697882
- [Derived] Jayalath VH, de Souza RJ, Ha V, Mirrahimi A, Blanco-Mejia S, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ, Sievenpiper JL. Sugar-sweetened beverage consumption and incident hypertension: a systematic review and meta-analysis of prospective cohorts. Am J Clin Nutr. 2015 Oct;102(4):914-21. doi: 10.3945/ajcn.115.107243. Epub 2015 Aug 12. PMID 26269365